CLINICAL TRIAL: NCT07241273
Title: SPECT-CT Guided ELEctive Contralateral Neck Treatment in Lateralized Oropharyngeal Cancer: A Phase II Trial
Brief Title: SPECT-CT Guided ELEctive Contralateral Neck Treatment in Lateralized Oropharyngeal Cancer
Acronym: SELECT-FR
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: UNICANCER (Other)
Collaborators: National Cancer Institute, France (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UC-RAD-2506; 2025-A00913-46 (Other: ANSM)
Record Dates: First submitted 2025-11-14; First posted 2025-11-21 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-10

CONDITIONS: Oropharyngeal Squamous Cell Carcinoma; Oropharyngeal Cancers; Oropharyngeal Carcinoma; Head and Neck; Head and Neck Cancer; Head and Neck Cancers
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Oropharyngeal Neoplasms; Head and Neck Neoplasms

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ipsilateral neck radiotherapy & SPECT-CT guided contralateral neck radiotherapy (Experimental): Radiotherapy of ipsilateral neck nodes & Radiotherapy of the contralateral neck nodes guided by SPECT-CT
  Interventions: Other: Lymphatic mapping with SPECT-CT; Radiation: Ipsilateral neck radiotherapy & SPECT-CT guided contralateral neck radiotherapy
- Bilateral neck radiotherapy (Active Comparator): Radiotherapy of nodes on both sides of the neck
  Interventions: Radiation: Bilateral neck radiotherapy

INTERVENTIONS:
Other: Lymphatic mapping with SPECT-CT — Lymphatic mapping with SPECT-CT
  Arms: Ipsilateral neck radiotherapy & SPECT-CT guided contralateral neck radiotherapy
Radiation: Bilateral neck radiotherapy — Patients will receive definitive radiotherapy to the primary tumour and bilateral neck nodes.
  Arms: Bilateral neck radiotherapy
Radiation: Ipsilateral neck radiotherapy & SPECT-CT guided contralateral neck radiotherapy — Patients will receive definitive radiotherapy to the primary tumour and ipsilateral neck nodes while radiotherapy to the contralateral neck nodes will be guided by lymphatic mapping with SPECT-CT.
  Arms: Ipsilateral neck radiotherapy & SPECT-CT guided contralateral neck radiotherapy

SUMMARY:
Oropharyngeal cancer (OPC) is the most common type of head and neck cancer. The current standard treatment for this cancer is radiotherapy (RT) of the tumour and lymph nodes of both sides of the neck, combined with concurrent chemotherapy for advanced stages. Even though a small proportion of patients with this cancer have involvement of the lymph nodes of the neck on the opposite side of the tumour (contralateral involvement) or involvement of the lymph nodes on both sides of the neck (bilateral involvement), bilateral radiotherapy is performed due to the risk of contralateral microscopic involvement, which is invisible on imaging and clinical examination. Bilateral radiotherapy causes more adverse events, leading to a decrease in quality of life.

Lymphatic mapping using Single Photon Emission Computed Tomography-Computed Tomography (SPECT-CT) imaging is a technique that visualises the lymphatic drainage of the tumour and thus determines whether radiotherapy should be delivered unilaterally or bilaterally to the lymph nodes. This technique would therefore reduce adverse events and improve quality of life, while maintaining the efficacy of radiotherapy.

The goal of the clinical trial SELECT-FR is to investigate if the efficacy of a lymphatic drainage mapping with a SPECT-CT-guided approach is acceptable in terms of two-year Disease Free Survival (DFS) rate in patients with lateralized OPC.

DETAILED DESCRIPTION:
SELECT-FR is a national, randomized, phase II, non-comparative trial.

Patients aged 18 or over, with lateralized oropharyngeal squamous cell carcinoma (tonsil, soft palate, pharyngeal wall or tongue base) not involving or crossing midline, Human Papilloma Virus (HPV) positive or negative, T1-T3 with no contralateral nodes or nodes > 6 cm on Computed Tomography (CT), Magnetic Resonance Imaging (MRI) or Positron Emission Tomography-Computed Tomography (PET-CT).

Eligible subjects will be randomized at a 1:1 ratio into the experimental and control arms.

* Experimental arm: Patients will receive definitive RT to the primary tumour and ipsilateral neck nodes, while contralateral neck RT treatment will be guided by lymphatic mapping with SPECT-CT.
* Control arm: Patients will receive definitive RT to the primary tumour and bilateral neck nodes (Note: candidates for standard unilateral neck RT are not eligible).

Randomization will be stratified by the following factors:

* Anatomical location of primary tumour: lateral vs. intermediate vs. medial.
* HPV status (p16 immunohistochemistry) and smoking status: p16 positive ≤ 10 pack year vs. p16 positive > 10 pack year vs. p16 negative any.
* Extent of disease: limited vs. other:

  * p16 positive: limited [T1-T2, N0-N1 (single node < 3cm without radiologic extranodal extension)] vs. other.
  * p16 negative: limited [T1-T2, N0-N1 (without radiologic extranodal extension)] vs. other.
* Use of concurrent systemic therapy: yes vs. no.

In both arms, time from randomization to initiation of RT will be no longer than 6 weeks. Patients will receive RT with or without standard concurrent chemotherapy in either standard fractionation (7 weeks) or altered fractionation (6 weeks).

In both arms, all patients will be followed by local investigator as follow:

* Treatment period: every week.
* Follow-up period: every 3 months until 24 months after treatment and then every 6 months until 36 months after treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have signed a written informed consent form prior to any trial specific procedures.
2. Patients with histologically confirmed T1-T3 M0 lateralized OPC (tonsil, soft palate, pharyngeal wall or base of tongue) not involving or crossing midline. Nodal disease may include no node or single or multiple ipsilateral lymph nodes (largest should be equal or less than 6 cm in maximum diameter) without contralateral nodes involved. For HPV-positive patients, this includes N0-N1. For HPV-negative patients, this includes N0-N2b. Patients with radiologic extranodal extension without clinical signs of extranodal extension (skin invasion, deep nodal fixation, and/or clinical signs of cranial nerve or brachial plexus invasion) will be eligible for participation.
3. HPV-positive or -negative (by p16 immunohistochemistry). Tumours will be classified as p16 at local sites based on greater than 70% strong diffuse nuclear or nuclear and cytoplasmic staining.
4. Planned definitive bilateral neck radiotherapy with or without concurrent chemotherapy.
5. Patients ≥ 18 years old.
6. ECOG Performance Status 0-1.
7. The following radiological investigations must have been done within 8 weeks before randomization:

   * CT or MRI of the neck (with head imaging as indicated);
   * PET-CT scan;
   * Chest CT scan.
8. Patients who receive a concomitant chemoradiotherapy (cCRT) should have adequate organ and bone marrow function including the following:

   * Hematological function (absolute neutrophil count ≥ 1.5 x10⁹/L, platelets ≥ 100 x10⁹/L, hemoglobin ≥ 9 g/dL) measured before cCRT.
   * Renal function (creatinine clearance ≥ 50 mL/min per Cockcroft and Gault formula) measured before cCRT.
   * Hepatic function (total bilirubin < 1.5 ULN, Aspartate aminotransferase (AST) and Alanine aminotransferase (ALT) < 2.5 ULN, Alkaline phosphatase < 2.5 ULN) measured before cCRT.
9. Women/men of childbearing potential must have agreed to use a highly effective contraceptive method up to 90 days after completing radiotherapy.

   Women of childbearing potential must have a negative pregnancy test before the beginning of the trial.
10. Treating surgeon must confirm that the patient is a candidate to undergo injection procedure for lymphatic mapping in either the nuclear medicine, ambulatory clinic, or operating room setting.
11. Patient is willing and able to comply with the protocol for the duration of the trial including undergoing treatment and scheduled visits, and examinations including follow-up.
12. Patients affiliated to (or beneficiary from) the French social security system.
13. Patients with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial.

Exclusion Criteria:

1. Patients with T1-T2 cancers isolated to the tonsil fossa (i.e., without any soft palate, tongue base, posterior pharyngeal wall or posterior tonsil pillar involvement) with no involved lymph nodes or with a single ipsilateral node < 3 cm without extranodal extension.
2. Patients with tonsil or tongue base primary squamous cell carcinoma who have previously undergone diagnostic palatine or lingual tonsillectomy with either complete excision or with no clinically apparent residual disease are excluded. However, patients who have had previous deep biopsies or partial excisions with clinically evaluable disease are still eligible.
3. Previous head and neck cancer or multiple synchronous primary head and neck cancers.
4. Previous induction or neo-adjuvant chemotherapy.
5. Previous radiation therapy to the head and neck or comprehensive neck dissection of at least 3 levels on either side (due to potential for disrupted lymphatic channels and drainage pathways). Patients who have had excisional biopsies of involved lymph nodes are, however, still eligible.
6. Previous radiotracer allergy. Contraindication in patients with history of hypersensitivity to human albumin-containing products.
7. Patients with severe, active co-morbidity including any of the following:

   * Chronic Obstructive Pulmonary Disease or other pulmonary illness requiring hospitalization within 30 days of registration.
   * Unstable angina and/or congestive heart failure requiring hospitalization within the 30 days of registration.
   * Acute myocardial infarction within 30 days of study registration.
   * Diseases precluding RT (e.g., scleroderma).
8. Presence of any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule, as assessed by the investigator.
9. Pregnant or breastfeeding women.
10. Patient enrolled in another therapeutic trial within 30 days of registration.
11. Persons deprived of their liberty or under protective custody or guardianship.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2030-04 (Estimated); Study Completion 2031-04 (Estimated)

PRIMARY OUTCOMES:
Two-years Disease Free Survival (DFS) rate | At 2 years after treatment
  The primary endpoint is 2 year-Disease-Free Survival rate (2y-DFS) defined as patients free of disease at two years. Patients without any event before 2 years will be considered as success, patients lost to follow-up before 2 years will be considered as failure.

SECONDARY OUTCOMES:
Disease free survival | From randomization to any of the following events: local, regional, or distant recurrence or death from any cause, up to 3 years after treatment.
  Disease-free survival (DFS) is defined as time from randomization to the date of first record of any of the following events including local, regional, or distant recurrence or death from any cause. DFS will be censored on the date of last visit with disease assessment.
Overall survival (OS) | From randomization to the date of death from any cause, up to 3 years after treatment.
  Overall survival (OS) is defined as the time from the date of randomization to the date of death from any cause. The follow-up of subjects still alive will be censored at the date of last visit/contact.
Isolated Contralateral Neck Failure (iCNF) | From randomization to the date of iCNF, up to 3 years after treatment.
  Isolated Contralateral Neck Failure (iCNF) is defined as the time from the date of randomization to the date of iCNF. Local ipsilateral neck failure, or distant failure diagnosed concurrently with iCNF or before are not considered events of interest but as competing risks events in the analysis of this endpoint. Subjects without any of the listed events (i.e. events of interest or competing risks events) are censored at the date of the most recent follow-up examination.
Local-regional failure (LRF) | From randomization to the date of any local or regional failure, up to 3 years after treatment.
  Local-regional failure (LRF) is defined as the time from the date of randomization to the date of any local or regional failure. Distant recurrence/progression diagnosed before local or regional failure are not considered events of interest, but as competing risks events in the analysis of this endpoint. Subjects without any of the listed events (i.e. events of interest or competing risks events) are censored at the date of the most recent follow-up examination.
Distant metastases (DM) | From randomization until clear evidence of distant metastasis, up to 3 years after treatment.
  Distant metastases (DM) are defined as clear evidence of distant metastases in the lung, bone, brain, liver or other distant sites. Biopsy is recommended where possible according to local practices. Distant sites can be evaluated by CT scans or PET-CT. Distant metastasis free survival is defined as the time from the date of randomization to the date of distant metastases. All other events are not considered events of interest, but as competing risks events in the analysis of this endpoint.
Incidence and Severity of Treatment-Related Adverse Events | Throughout study completion, up to 3 years after treatment.
  Toxicities will be measured using the National Cancer Institute-Common Terminology Criteria for Adverse Events version 5 (NCI-CTCAE v5.0). The NCI-CTCAE is a descriptive terminology which can be used for Adverse Event (AE) reporting and it is widely accepted in the community of oncology research as the leading rating scale for adverse events. A grading (severity) scale is provided for each AE term. This scale is divided into 5 grades (1 = "mild", 2 = "moderate", 3 = "severe", 4 = "life-threatening", and 5 = "death"). Toxicities will be measured by the investigator weekly during Radiotherapy (RT), at 1 month and 3 months after completion of RT to assess acute toxicities and then at each follow up visit following completion of RT to assess late toxicities until 36 months post RT.
Incidence and Severity of Treatment-Related Adverse Events reported by patients (using items of PRO-CTCAE) | Throughout study completion, up to 2 years after treatment.
  Patient reported toxicities will be evaluated using selected items of the validated Patient-Reported Outcome-Common Terminology Criteria for Adverse Events (PRO-CTCAE). It is recognized that clinician-reported adverse events (AEs) may substantially under-report the incidence and severity of symptoms occurring as a consequence of treatment. In response to this awareness, the NCI has developed a set of patient-reported items (called PRO-CTCAE) that complement the CTCAE and capture the patient's perspective on the subjective aspects of adverse events. PRO-CTCAE H&N information will complement the clinician CTCAE reporting. A collection of 15 specific PRO-CTCAE Head & Neck (H&N) items is proposed. Patient reported toxicities will be evaluated at baseline, end of treatment, 12, and 24 months after the end of treatment.
Gastrostomy tube usage | Throughout study completion, up to 3 years after treatment.
  Gastrostomy tube usage will be assessed for the presence of a gastrostomy tube as well as usage of the gastrostomy tube at each visit until tube removal.

CONTACTS AND LOCATIONS:
Overall Officials: Sébastien THUREAU, MD, Study Chair — Centre Henri Becquerel
Locations (12):
- France (12):
  - CHU Brest, Brest
  - Centre François Baclesse, Caen
  - CHU Caen, Caen
  - Centre Georges François Leclerc, Dijon
  - Centre de Radiothérapie Guillaume Le Conquérant, Le Havre
  - Centre Oscar Lambret, Lille
  - Institut Régional du Cancer de Montpellier, Montpellier
  - Hôpital Tenon, Paris
  - Centre Henri Becquerel, Rouen
  - Hôpitaux Universitaires de Strasbourg - Hôpital de Hautepierre, Strasbourg
  - Institut de Cancérologie Strasbourg Europe, Strasbourg
  - CHRU Tours - Hôpital Bretonneau, Tours

IPD SHARING:
Plan to Share IPD: No